CLINICAL TRIAL: NCT04721821
Title: Comparative Effectiveness of Tumor Necrosis Factor (TNF) Inhibitors and Tofacitinib, Overall, by Line of Therapy and by Combination Therapy
Brief Title: Comparative Effectiveness Of Tumor Necrosis Factor Inhibitors And Tofacitinib Use In Earlier Lines Of Therapy And Use As Monotherapy.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921389
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Arthritis Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Rheumatoid Arthritis (RA)
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Patients who received Tofacitinib for RA

SUMMARY:
This study is to investigate if there has been a shift in treatment with tofacitinib, assessing real world patient data and entered in the Corrona registry between 2016 and 2020.

ELIGIBILITY:
Inclusion Criteria:

* RA patients in Corrona initiating tofacitinib or a TNF biologic (adalimumab, etanercept, infliximab, golimumab, certolizumab pegol) after 06 November 2012 (market approval of Tofacitinib) during follow-up in Corrona with no prior use of tofacitinib. Only the patient's first initiation after 06 November 2012 will be included in the analysis
* Have a 6 and / or 12-month follow-up visit (with +/- 2 month window)
* Have Clinical Disease Activity Index (CDAI) measures at baseline and at the follow-up visit

Exclusion Criteria:

* Patients who have not failed methotrexate (MTX) or another csDMARD (ie 1st line initiators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected from the Corrona RA Registry. The Corrona RA Registry is a prospective, multicenter, observational disease-based registry.
Sampling Method: Non-Probability Sample
Enrollment: 7807 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with rheumatoid arthritis (RA), enrolled in Corrona RA registry, initiated tofacitinib or tumor necrosis factor inhibitors (TNFis) on or after 06-November-2012, after failure with conventional synthetic disease modifying antirheumatic drugs (csDMARDs) treatment, were included.
Pre-assignment Details: Data was collected retrospectively for observation period from 06-November-2012 to 28-Feb-2021 (approximately 8.3 years). Data from eligible participants for aforesaid observation period were retrieved and observed in this retrospective study from 22-January-2021 to 29-November-2021 (approximately 10 months).
Groups:
- Tofacitinib (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
- TNFis (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
- Tofacitinib (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
- TNFis (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
Period: Overall Study
Arm/Group | Tofacitinib (6-Month Follow-up) | TNFis (6-Month Follow-up) | Tofacitinib (12-Month Follow-up) | TNFis (12-Month Follow-up)
Started | 989 | 3337 | 805 | 2676
Completed | 989 | 3337 | 805 | 2676
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were observed in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib (6-Month Follow-up) | TNFis (6-Month Follow-up) | Tofacitinib (12-Month Follow-up) | TNFis (12-Month Follow-up) | Total
Number analyzed (Participants) | 989 | 3337 | 805 | 2676 | 7807
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: "Number Analyzed" refers to those participants whose data was available and is reported. Data for remaining participants was missing and not reported.
  Years
    number analyzed (Participants) | 987 | 3334 | 803 | 2671 | 7795
    (all) | 60.5 (11.8) | 58.4 (12.8) | 59.9 (11.9) | 58.9 (12.6) | 59.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: "Number Analyzed" refers to those participants whose data was available and is reported. Data for remaining participants was missing and not reported.
  Participants
    number analyzed (Participants) | 987 | 3337 | 803 | 2674 | 7801
    Female | 804 | 2634 | 651 | 2094 | 6183
    Male | 183 | 703 | 152 | 580 | 1618
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 846 | 2,716 | 697 | 2199 | 6458
  Hispanic | 67 | 272 | 53 | 192 | 584
  Black | 42 | 212 | 30 | 167 | 451
  Asian | 6 | 55 | 6 | 40 | 107
  Other | 13 | 50 | 5 | 44 | 112
  Missing | 15 | 32 | 14 | 34 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Low Disease Activity (LDA) Based on Clinical Disease Activity Index (CDAI) at Month 6: Tofacitinib Overall Versus TNFis Overall
Description: CDAI was a simplified index for assessing the disease activity comprising of the swollen joint counts (SJC), tender/painful joint counts (TJC), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA). CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment range from 0 to 28, higher scores meant worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 centimeter (cm) visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Achievement of LDA was defined by CDAI less than or equal to (<=)10 in participants with moderate or high disease activity CDAI greater than (>) 10 at baseline. Propensity score method was used for analysis of the outcome measure.
Time Frame: Month 6 visit post initiation of Tofacitinib or TNFis, during observation period from 06-November-2012 to 28-Feb-2021 (approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: Eligible participants whose data were observed in this study. Here for this outcome measure analysis, "Overall Number of Participants Analyzed" refers to evaluable participants who were matched using propensity score method for respective reporting arms and had moderate or high disease activity (CDAI>10) at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Overall (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as monotherapy or combination therapy with csDMARDs after 06-November-2012 and had at least 6- month follow-up post initiation, were included in this reporting arm.
- TNFis Overall (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as monotherapy or combination therapy with csDMARDs after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up)
Number analyzed (Participants) | 502 | 513
Participants | 129 | 140
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.82 to 1.44]

2. Primary Outcome: Number of Participants Who Achieved LDA Based on CDAI at Month 6: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: CDAI was a simplified index for assessing the disease activity comprising of the SJC, TJC, PtGA and PGA. CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment, range from 0 to 28, higher scores meant worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 cm visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Achievement of LDA was defined by CDAI <=10 in participants with moderate or high disease activity CDAI>10 at baseline. Propensity score method was used for analysis of the outcome measure.
Time Frame: Month 6 visit post initiation of Tofacitinib during observation period from 06-November-2012 to 28-Feb-2021 (approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: Eligible participants whose data were observed in this study. Here for this outcome measure analysis, "Overall Number of Participants Analyzed" refers to evaluable participants who were matched using propensity score method for respective reporting arms and had moderate or high disease activity CDAI >10 at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Monotherapy (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as monotherapy after 06-November-2012 and had at least 6- month follow-up post initiation, were included in this reporting arm.
- Tofacitinib Combination Therapy (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as combination therapy with csDMARDs after 06-November-2012 and had at least 6- month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up)
Number analyzed (Participants) | 228 | 231
Participants | 66 | 48
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.44 to 1.16]

3. Primary Outcome: Number of Participants Who Achieved LDA Based on CDAI at Month 6: TNFi Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 2
Time Frame: Month 6 visit post initiation of TNFis, during observation period from 06-November-2012 to 28-Feb-2021 (approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- TNFis Monotherapy (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as monotherapy after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
- TNFis Combination Therapy (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as combination therapy with csDMARDs after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up)
Number analyzed (Participants) | 469 | 438
Participants | 166 | 154
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.73 to 1.27]

4. Primary Outcome: Number of Participants Who Achieved LDA Based on CDAI at Month 6: Tofacitinib Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up)
Number analyzed (Participants) | 223 | 222
Participants | 59 | 68
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.79 to 1.88]

5. Primary Outcome: Number of Participants Who Achieved LDA Based on CDAI at Month 6: Tofacitinib Combination Therapy Versus TNFis Combination Therapy
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- TNFis Combination Therapy (6 Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as combination therapy with csDMARDs after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6 Month Follow-up)
Number analyzed (Participants) | 310 | 301
Participants | 82 | 82
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6 Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.79 to 1.67]

6. Primary Outcome: Number of Participants Who Achieved LDA Based on CDAI at Month 12: Tofacitinib Overall Versus TNFis Overall
Description: as for outcome 2
Time Frame: Month 12 visit post initiation of Tofacitinib or TNFis, during observation period from 06-November-2012 to 28-Feb-2021 (approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Overall (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as monotherapy or combination therapy with csDMARDs after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
- TNFis Overall (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as monotherapy or combination therapy with csDMARDs after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 419 | 417
Participants | 104 | 127
Statistical Analysis 1: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.94 to 1.76]

7. Primary Outcome: Number of Participants Who Achieved LDA Based on CDAI at Month 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: as for outcome 2
Time Frame: Month 12 visit post initiation of Tofacitinib during observation period from 06-November-2012 to 28-Feb-2021 (approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Monotherapy (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as monotherapy after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
- Tofacitinib Combination Therapy (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as combination therapy with csDMARDs after 06-November-2012 and had at least 12- month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 180 | 176
Participants | 44 | 48
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.70 to 1.89]

8. Primary Outcome: Number of Participants Who Achieved LDA Based on CDAI at Month 12: TNFis Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 2
Time Frame: Month 12 visit post initiation of TNFis, during observation period from 06-November-2012 to 28-Feb-2021 (approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- TNFis Monotherapy (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as monotherapy after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
- TNFis Combination Therapy (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as combination therapy with csDMARDs after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
Arm/Group | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 362 | 356
Participants | 123 | 129
Statistical Analysis 1: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.69 to 1.32]

9. Primary Outcome: Number of Participants Who Achieved LDA Based on CDAI at Month 12: Tofacitinib Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 2
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- TNFis Combination Therapy (12- Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as combination therapy with csDMARDs after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12- Month Follow-up)
Number analyzed (Participants) | 160 | 165
Participants | 40 | 52
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12- Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.81 to 2.16]

10. Primary Outcome: Number of Participants Who Achieved LDA Based on CDAI at Month 12: Tofacitinib Combination Therapy Versus TNFis Combination Therapy
Description: as for outcome 2
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 234 | 240
Participants | 57 | 67
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Test type: Superiority; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.81 to 1.87]

11. Secondary Outcome: Number of Participants Who Achieved Remission Based on CDAI at Month 6 and 12: Tofacitinib Overall Versus TNFis Overall
Description: CDAI was a simplified index for assessing the disease activity comprising of the SJC, TJC, PtGA and PGA. CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment, range from 0 to 28, higher scores meant worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 cm visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Achievement of remission was defined by CDAI (<=2.8) in those participants with LDA, moderate or high disease activity (CDAI >2.8) at baseline. Propensity score method was used for analysis of the outcome measure.
Time Frame: Months 6 and 12 visit(for respective arms)post initiation of Tofacitinib or TNFis,during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years);data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: Eligible participants whose data were observed in this study. Here for this outcome measure analysis, "Overall Number of Participants Analyzed" refers to evaluable participants who were matched using propensity score method for respective reporting arms and had LDA, moderate or high disease activity (CDAI >2.8) at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 686 | 680 | 572 | 565
Participants | 61 | 71 | 53 | 61
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.80 to 1.66]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.75 to 1.65]

12. Secondary Outcome: Number of Participants Who Achieved Remission Based on CDAI at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: as for outcome 11
Time Frame: Months 6 and 12 visit(for respective arms)post initiation of Tofacitinib during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years);data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Monotherapy (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
- Tofacitinib Monotherapy (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
- Tofacitinib Combination Therapy (12-Month Follow-up: Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as combination therapy with csDMARDs after 06-November-2012 and had at least 12- month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up
Number analyzed (Participants) | 317 | 311 | 259 | 251
Participants | 29 | 23 | 23 | 24
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.57 to 1.99]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up; Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.49 to 1.75]

13. Secondary Outcome: Number of Participants Who Achieved Remission Based on CDAI at Month 6 and 12: TNFis Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 11
Time Frame: Months 6 and 12 visit(for respective arms)post initiation of TNFis, during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years);data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 606 | 604 | 474 | 485
Participants | 69 | 78 | 55 | 56
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.79 to 1.58]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.60 to 1.35]

14. Secondary Outcome: Number of Participants Who Achieved Remission Based on CDAI at Month 6 and 12: Tofacitinib Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Monotherapy (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as monotherapy after 06-November-2012 and had at least 12- month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 315 | 316 | 230 | 236
Participants | 28 | 36 | 20 | 30
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.77 to 2.29]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.82 to 2.71]

15. Secondary Outcome: Number of Participants Who Achieved Remission Based on CDAI at Month 6 and 12: Tofacitinib Combination Therapy Versus TNFis Combination Therapy
Description: as for outcome 11
Time Frame: Month 6 and 12 visit(for respective arms)post initiation of Tofacitinib or TNFis, during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years);data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- TNFis Combination Therapy (12 Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as combination therapy with csDMARDs after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12 Month Follow-up)
Number analyzed (Participants) | 414 | 412 | 319 | 317
Participants | 34 | 41 | 26 | 23
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.81 to 2.24]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12 Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.50 to 1.62]

16. Secondary Outcome: Change From Baseline in CDAI 0-76 at Month 6 and 12: Tofacitinib Overall Versus TNFis Overall
Description: CDAI was a simplified index for assessing the disease activity comprising of the SJC, TJC, PtGA and PGA. CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment, range from 0 to 28, higher scores meant worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 cm visual analog scale; higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Propensity score method was used for analysis of the outcome measure.
Time Frame: Baseline, Months 6 and 12 visit (for respective arms) post initiation of Tofacitinib or TNFis, during observation period from 06-Nov-2012 to 28-Feb-2021 (approximately 8.3 years);data collected and studied from 22-Jan-2021 to 29-Nov-2021 in this study
Population: Eligible participants whose data were observed in this study. Here for this outcome measure analysis, "Overall Number of Participants Analyzed" refers to evaluable participants who were matched using propensity score method for respective reporting arms.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- TNFis Overall (6 Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as monotherapy or combination therapy with csDMARDs after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6 Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 735 | 735 | 611 | 611
Units on a scale | -3.85 (12.71) | -3.98 (12.64) | -3.29 (13.28) | -4.39 (11.82)
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6 Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.88 to 1.31]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Net) = -1.50, 95% CI 2-sided [-2.73 to -0.27]

17. Secondary Outcome: Change From Baseline in CDAI 0-76 at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: as for outcome 16
Time Frame: Baseline,Months 6 and 12 visit(for respective arms)post initiation of Tofacitinib during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years);data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Tofacitinib Monotherapy (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as monotherapy after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
- Tofacitinib Combination Therapy (12-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as combination therapy with csDMARDs after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 345 | 345 | 277 | 277
Units on a scale | -3.43 (12.77) | -2.66 (12.59) | -3.30 (13.68) | -2.31 (12.23)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Median Difference (Net) = 0.39, 95% CI 2-sided [-1.24 to 2.02]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Median Difference (Net) = 0.96, 95% CI 2-sided [-0.92 to 2.84]

18. Secondary Outcome: Change From Baseline in CDAI 0-76 at Month 6 and 12: TNFis Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 16
Time Frame: Baseline, Months 6 and 12 visit(for respective arms)post initiation of TNFis, during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years);data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 670 | 670 | 536 | 536
Units on a scale | -4.39 (12.32) | -4.36 (11.82) | -5.07 (12.08) | -3.49 (11.76)
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Net) = -0.56, 95% CI 2-sided [-1.68 to 0.56]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Net) = 0.74, 95% CI 2-sided [-0.51 to 1.99]

19. Secondary Outcome: Change From Baseline in CDAI 0-76 at Month 6 and 12: Tofacitinib Monotherapy vs TNFis Combination Therapy
Description: as for outcome 16
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 343 | 343 | 246 | 246
Units on a scale | -3.26 (12.68) | -3.66 (12.41) | -3.33 (13.51) | -4.39 (10.85)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Net) = -1.11, 95% CI 2-sided [-2.66 to 0.45]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Net) = -1.73, 95% CI 2-sided [-3.52 to 0.05]

20. Secondary Outcome: Change From Baseline in CDAI 0-76 at Month 6 and 12: Tofacitinib Combination Therapy vs TNFis Combination Therapy
Description: as for outcome 16
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 443 | 443 | 344 | 344
Units on a scale | -3.92 (13.20) | -4.53 (11.94) | -3.28 (12.59) | -4.29 (12.23)
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Net) = -0.93, 95% CI 2-sided [-2.30 to 0.44]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Net) = -0.99, 95% CI 2-sided [-2.60 to 0.62]

21. Secondary Outcome: Number of Participants With Modified American College of Rheumatology (mACR) 20/50/70 at Month 6 and 12: Tofacitinib Overall Versus TNFis Overall
Description: mACR 20/50/70 response was defined as response greater than or equal to( >=) 20 percent (%), 50%, or 70% improvement in tender and swollen joint count and 20%, 50% or 70% improvement respectively in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the modified Health Assessment Questionnaire (mHAQ) [scored from 0 to 3, higher scores indicated worsening of function]. Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 731 | 730 | 608 | 602
Participants
  mACR 20 | 138 | 143 | 114 | 109
  mACR 50 | 73 | 87 | 52 | 63
  mACR 70 | 33 | 32 | 22 | 33
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.80 to 1.35]
Statistical Analysis 2: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.86 to 1.67]
Statistical Analysis 3: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.57 to 1.54]
Statistical Analysis 4: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.77 to 1.41]
Statistical Analysis 5: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.89 to 1.95]
Statistical Analysis 6: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.85 to 2.60]

22. Secondary Outcome: Number of Participants With MACR 20/50/70 at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: mACR 20/50/70 response was defined as response >= 20%, 50%, or 70% improvement in tender and swollen joint count and 20%, 50% or 70% improvement respectively in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsening of pain); 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsening of condition); 4) self-assessed disability index of the mHAQ (scored from 0 to 3, higher scores indicated worsening of function). Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 12
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Combination Therapy (6-Month Follow-up)): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as combination therapy with csDMARDs after 06-November-2012 and had at least 6- month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up)) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 333 | 328 | 272 | 267
Participants
  mACR 20 | 63 | 56 | 46 | 43
  mACR 50 | 38 | 25 | 20 | 19
  mACR 70 | 15 | 10 | 12 | 8
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up)); Month 6 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.59 to 1.34]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up)); Month 6 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.39 to 1.15]
Statistical Analysis 3: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up)); Month 6 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.34 to 1.83]
Statistical Analysis 4: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.56 to 1.42]
Statistical Analysis 5: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.46 to 1.80]
Statistical Analysis 6: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.19 to 1.48]

23. Secondary Outcome: Number of Participants With MACR 20/50/70 at Month 6 and 12: TNFis Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 22
Time Frame: as for outcome 13
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 666 | 663 | 531 | 533
Participants
  mACR 20 | 137 | 151 | 111 | 107
  mACR 50 | 90 | 85 | 59 | 59
  mACR 70 | 47 | 35 | 34 | 26
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.86 to 1.45]
Statistical Analysis 2: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.67 to 1.26]
Statistical Analysis 3: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.44 to 1.09]
Statistical Analysis 4: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.74 to 1.38]
Statistical Analysis 5: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.69 to 1.52]
Statistical Analysis 6: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.46 to 1.33]

24. Secondary Outcome: Number of Participants With MACR 20/50/70 at Month 6 and 12: Tofacitinib Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 22
Time Frame: as for outcome 15
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Groups:
- TNFis Combination Therapy (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
- Tofacitinib Monotherapy (12 Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as monotherapy after 06-November-2012 and had at least 12- month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12 Month Follow-up) | TNFis Combination Therapy (12 Month Follow-up)
Number analyzed (Participants) | 338 | 340 | 244 | 244
Participants
  mACR 20 | 66 | 66 | 42 | 33
  mACR 50 | 36 | 37 | 21 | 19
  mACR 70 | 13 | 12 | 12 | 9
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.78 to 1.77]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.71 to 1.95]
Statistical Analysis 3: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.45 to 2.39]
Statistical Analysis 4: Comparison: Tofacitinib Monotherapy (12 Month Follow-up) vs TNFis Combination Therapy (12 Month Follow-up); Month 12 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.50 to 1.40]
Statistical Analysis 5: Comparison: Tofacitinib Monotherapy (12 Month Follow-up) vs TNFis Combination Therapy (12 Month Follow-up); Month 12 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.49 to 1.83]
Statistical Analysis 6: Comparison: Tofacitinib Monotherapy (12 Month Follow-up) vs TNFis Combination Therapy (12 Month Follow-up); Month 12 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.33 to 1.95]

25. Secondary Outcome: Number of Participants With MACR 20/50/70 at Month 6 and 12: Tofacitinib Combination Therapy Versus TNFis Combination Therapy
Description: as for outcome 22
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Combination Therapy (6-Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as combination therapy with csDMARDs after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 442 | 439 | 343 | 341
Participants
  mACR 20 | 91 | 91 | 65 | 57
  mACR 50 | 47 | 39 | 30 | 32
  mACR 70 | 24 | 16 | 10 | 14
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.76 to 1.49]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.55 to 1.37]
Statistical Analysis 3: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.32 to 1.20]
Statistical Analysis 4: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 20; Test type: Superiority; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.59 to 1.30]
Statistical Analysis 5: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 50; Test type: Superiority; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.65 to 1.86]
Statistical Analysis 6: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis: mACR 70; Test type: Superiority; Odds Ratio (OR) = 1.43, 95% CI [0.62 to 3.28]

26. Secondary Outcome: Number of Participants Who Achieved LDA Based on Disease Activity Score (DAS 28) Erythrocyte Sedimentation Rate (ESR) at Month 6 and 12: Tofacitinib Overall Versus TNFis Overall
Description: DAS28 ESR was calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, ESR (millimeters per hour [mm/hour]) and participant's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated high disease activity). DAS 28 ESR =0.56*sqrt (PJC28) + 0.28*sqrt (SJC28) + 0.70*In (ESR) + 0.014*PtGA; ln = natural logarithm, sqrt = square root of. DAS28 ESR <= 3.2 = low disease activity, DAS28 ESR > 3.2 and <=5.1 = moderate and >5.1 = high disease activity. Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 11
Population: Eligible participants whose data were observed in this study. Here for this outcome measure analysis, "Overall Number of Participants Analyzed" refers to evaluable participants who were matched using propensity score method for respective reporting arms and DAS28 ESR >3.2 at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 314 | 279 | 265 | 232
Participants | 54 | 64 | 44 | 40
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.94 to 2.15]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.68 to 1.84]

27. Secondary Outcome: Number of Participants Who Achieved LDA Based on DAS 28 ESR at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: DAS28 ESR was calculated from the number of SJC and PJC using the 28 joints count, ESR (mm/hour) and PGA of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated high disease activity). DAS 28 ESR =0.56*sqrt (PJC28) + 0.28*sqrt (SJC28) + 0.70*In (ESR) + 0.014*PtGA; ln = natural logarithm, sqrt = square root of. DAS28 ESR <= 3.2 = low disease activity, DAS28 ESR > 3.2 and <=5.1 = moderate and >5.1 = high disease activity. Propensity score method was used for analysis of the outcome measure.
Time Frame: Months 6 and 12 visit (for respective arms)post initiation of Tofacitinib during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years);data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 131 | 149 | 112 | 108
Participants | 24 | 20 | 14 | 16
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.41 to 1.67]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.62 to 3.07]

28. Secondary Outcome: Number of Participants Who Achieved LDA Based on DAS 28 ESR at Month 6 and 12: TNFis Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 27
Time Frame: as for outcome 13
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12 Month Follow-up)
Number analyzed (Participants) | 255 | 236 | 204 | 205
Participants | 62 | 56 | 39 | 45
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.66 to 1.52]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12 Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.64 to 1.74]

29. Secondary Outcome: Number of Participants Who Achieved LDA Based on DAS 28 ESR at Month 6 and 12: Tofacitinib Monotherapy Versus TNFis Combination Therapy
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 129 | 129 | 95 | 88
Participants | 23 | 32 | 12 | 17
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.80 to 2.94]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.76 to 3.87]

30. Secondary Outcome: Number of Participants Who Achieved LDA Based on DAS 28 ESR at Month 6 and 12: Tofacitinib Combination Therapy vs TNFis Combination Therapy
Description: as for outcome 27
Time Frame: as for outcome 11
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 201 | 167 | 151 | 143
Participants | 36 | 34 | 24 | 24
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.73 to 2.27]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.63 to 2.23]

31. Secondary Outcome: Health Assessment Questionnaire (HAQ) Score at Month 6 and 12: Tofacitinib Overall Versus TNFis Overall
Description: HAQ: self-reported, valid assessment of functional disability in RA. The 20-question instrument assessed ability of participants to perform daily activities in 8 functional areas: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. Eight items were rated on a 4-point Likert scale from 0 to 3, where 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning. Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 735 | 735 | 611 | 611
Units on a scale | 1.02 (0.71) | 1.06 (0.71) | 0.98 (0.73) | 1.05 (0.74)
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.06 to 0.04]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.01 to 0.09]

32. Secondary Outcome: HAQ Score at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: as for outcome 31
Time Frame: as for outcome 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 345 | 345 | 277 | 277
Units on a scale | 1.05 (0.72) | 1.10 (0.70) | 1.06 (0.74) | 1.04 (0.75)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.08 to 0.06]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Median Difference (Final Values) = -0.03, 95% CI 2-sided [-0.11 to 0.05]

33. Secondary Outcome: HAQ Score at Month 6 and 12: TNFi Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 31
Time Frame: as for outcome 13
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6 Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 670 | 670 | 536 | 536
Units on a scale | 0.92 (0.71) | 0.88 (0.70) | 0.95 (0.71) | 0.98 (0.73)
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6 Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.07 to 0.03]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.01, 95% CI 2-sided [-0.05 to 0.07]

34. Secondary Outcome: HAQ Score at Month 6 and 12: Tofacitinib Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 31
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12 Month Follow-up)
Number analyzed (Participants) | 343 | 343 | 246 | 246
Units on a scale | 0.98 (0.69) | 1.00 (0.67) | 1.01 (0.72) | 0.99 (0.73)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.06 to 0.07]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12 Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.12 to 0.06]

35. Secondary Outcome: HAQ Score at Month 6 and 12: Tofacitinib Combination Therapy Versus TNFi Combination Therapy
Description: as for outcome 31
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 443 | 443 | 344 | 344
Units on a scale | 1.04 (0.70) | 1.10 (0.73) | 0.99 (0.75) | 1.04 (0.76)
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.09 to 0.04]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.02, 95% CI 2-sided [-0.06 to 0.09]

36. Secondary Outcome: Number of Participants Who Achieved Minimally Clinically Important Difference (MCID) at Month 6 and 12: Tofacitinib Overall Versus TNFi Overall
Description: MCID improvement assessed based on HAQ. HAQ: self-reported, valid assessment of functional disability in RA. Assessed based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. Eight items were rated on a 4-point Likert scale from 0 to 3, where 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning. Achievement of MCID for the HAQ was defined as decrease in minimum of 0.22 units from baseline. Propensity score method was used for analysis of the outcome measure.
Time Frame: Months 6 and 12 visit (for respective arms) post initiation of Tofacitinib or TNFis, during observation period from 06-Nov-2012 to 28-Feb-2021 (approximately 8.3 years);data collected and studied from 22-Jan-2021 to 29-Nov-2021 in this study
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 614 | 618 | 507 | 504
Participants | 197 | 213 | 174 | 135
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.90 to 1.45]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.54 to 0.94]

37. Secondary Outcome: Number of Participants Who Achieved MCID at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: as for outcome 36
Time Frame: Months 6 and 12 visit (for respective arms) post initiation of Tofacitinib during observation period from 06-Nov-2012 to 28-Feb-2021 (approximately 8.3 years);data collected and studied from 22-Jan-2021 to 29-Nov-2021 in this study
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Combination Therapy (12- Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as combination therapy with csDMARDs after 06-November-2012 and had at least 12- month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12- Month Follow-up)
Number analyzed (Participants) | 269 | 278 | 226 | 221
Participants | 94 | 82 | 73 | 75
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.53 to 1.11]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12- Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.72 to 1.61]

38. Secondary Outcome: Number of Participants Who Achieved MCID at Month 6 and 12: TNFi Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 36
Time Frame: Baseline, Months 6 and 12 visit (for respective arms) post initiation of TNFis, during observation period from 06-Nov-2012 to 28-Feb-2021 (approximately 8.3 years);data collected and studied from 22-Jan-2021 to 29-Nov-2021 in this study
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 543 | 539 | 429 | 452
Participants | 202 | 197 | 129 | 143
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.73 to 1.21]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.77 to 1.39]

39. Secondary Outcome: Number of Participants Who Achieved MCID at Month 6 and 12: Tofacitinib Monotherapy vs TNFi Combination Therapy
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 269 | 286 | 199 | 201
Participants | 97 | 95 | 62 | 62
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.64 to 1.32]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.69 to 1.64]

40. Secondary Outcome: Number of Participants Who Achieved MCID at Month 6 and 12: Tofacitinib Combination Therapy vs TNFi Combination Therapy
Description: as for outcome 36
Time Frame: as for outcome 36
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Combination Therapy (6- Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib as combination therapy with csDMARDs after 06-November-2012 and had at least 6- month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib Combination Therapy (6- Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 379 | 381 | 290 | 281
Participants | 121 | 131 | 94 | 86
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6- Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.84 to 1.59]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.65 to 1.32]

41. Secondary Outcome: Modified Health Assessment Questionnaire (mHAQ) Score at Month 6 and 12: Tofacitinib Overall Versus TNFi Overall
Description: mHAQ is the modified version of HAQ which simplifies it from 20 questions to 8 questions, which assessed the ability to perform tasks due to rheumatoid arthritis. It comprised of 8 questions on 8 categories of daily living activities: dress/groom; arise; eat; grip; walk; hygiene; reach; and common activities over past week before specified time point. Eight items were rated on a 4-point Likert scale from 0 to 3, where 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score ranged from 0 to 3, where 0 = least difficulty and 3 = extreme difficulty, higher scores indicating worse functioning. Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 735 | 735 | 611 | 611
Units on a scale | 0.51 (0.50) | 0.53 (0.51) | 0.52 (0.54) | 0.53 (0.51)
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.03 to 0.04]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.04 to 0.05]

42. Secondary Outcome: mHAQ Score at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: as for outcome 41
Time Frame: as for outcome 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up)) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 345 | 345 | 277 | 277
Units on a scale | 0.55 (0.52) | 0.56 (0.50) | 0.57 (0.55) | 0.55 (0.52)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up)); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.05 to 0.05]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.07 to 0.06]

43. Secondary Outcome: mHAQ Score at Month 6 and 12: TNFi Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 41
Time Frame: as for outcome 13
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- TNFis Monotherapy (12-Month Follow-up: Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) as monotherapy after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 670 | 670 | 536 | 536
Units on a scale | 0.48 (0.48) | 0.44 (0.47) | 0.48 (0.47) | 0.49 (0.51)
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.06 to 0.02]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.04 to 0.04]

44. Secondary Outcome: mHAQ Score at Month 6 and 12: Tofacitinib Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 41
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 343 | 343 | 246 | 246
Units on a scale | 0.50 (0.48) | 0.50 (0.50) | 0.53 (0.52) | 0.49 (0.50)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.06 to 0.04]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.10 to 0.03]

45. Secondary Outcome: mHAQ Score at Month 6 and 12: Tofacitinib Combination Therapy Versus TNFi Combination Therapy
Description: as for outcome 41
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 443 | 443 | 344 | 344
Units on a scale | 0.51 (0.49) | 0.56 (0.54) | 0.51 (0.54) | 0.53 (0.53)
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.05 to 0.04]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.06 to 0.06]

46. Secondary Outcome: Pain Visual Analog Scale (VAS) at Month 6 and 12: Tofacitinib Overall Versus TNFi Overall
Description: Pain VAS was assessed using 100 millimeter (mm) horizontal line to rate pain. Score ranged from 0 mm to 100 mm; where, 0 = no pain and 100 = worst possible pain. Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 735 | 735 | 611 | 611
Millimeter | 43.61 (29.07) | 44.33 (28.80) | 43.22 (29.02) | 43.45 (29.22)
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-2.65 to 2.45]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-2.59 to 3.11]

47. Secondary Outcome: Pain VAS at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: Pain VAS was assessed using 100 mm horizontal line to rate pain. Score ranged from 0 mm to 100 mm; where, 0 = no pain and 100 = worst possible pain. Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 345 | 345 | 277 | 277
Millimeter | 43.99 (29.28) | 44.89 (28.54) | 46.91 (28.38) | 44.21 (28.90)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-2.71 to 4.38]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-5.12 to 2.95]

48. Secondary Outcome: Pain VAS at Month 6 and 12: TNFi Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 47
Time Frame: as for outcome 13
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 670 | 670 | 536 | 536
Millimeter | 42.70 (29.43) | 41.80 (28.60) | 42.74 (28.97) | 42.87 (29.33)
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-3.94 to 1.45]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-3.61 to 2.42]

49. Secondary Outcome: Pain VAS at Month 6 and 12: Tofacitinib Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 47
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 343 | 343 | 246 | 246
Millimeter | 43.56 (29.23) | 42.97 (27.64) | 46.11 (28.41) | 41.82 (28.53)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-4.39 to 3.05]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -4.84, 95% CI 2-sided [-9.19 to -0.48]

50. Secondary Outcome: Pain VAS at Month 6 and 12: Tofacitinib Combination Therapy vs TNFi Combination Therapy
Description: as for outcome 47
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 443 | 443 | 443 | 443
Millimeter | 43.62 (28.79) | 44.30 (28.80) | 43.13 (29.48) | 44.62 (29.08)
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-3.59 to 2.82]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-2.97 to 4.49]

51. Secondary Outcome: Number of Participants Who Experienced Mild Pain at Month 6 and 12: Tofacitinib Overall Versus TNFi Overall
Description: Pain VAS was assessed using 100 mm horizontal line to rate pain. Score ranged from 0 mm to 100 mm; where, 0 = no pain and 100 = worst possible pain. Participants who reported VAS <= 20 mm were categorized with mild pain and were reported in this outcome measure. Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 564 | 586 | 472 | 476
Participants | 98 | 102 | 79 | 79
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.73 to 1.34]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.66 to 1.34]

52. Secondary Outcome: Number of Participants Who Experienced Mild Pain at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: as for outcome 51
Time Frame: as for outcome 27
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 261 | 265 | 214 | 209
Participants | 43 | 42 | 30 | 27
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.62 to 1.73]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.50 to 1.60]

53. Secondary Outcome: Number of Participants Who Experienced Mild Pain at Month 6 and 12: TNFi Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 51
Time Frame: Months 6 and 12 visit (for respective arms) post initiation of TNFis, during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 524 | 520 | 409 | 428
Participants | 107 | 96 | 73 | 71
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.64 to 1.19]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.60 to 1.26]

54. Secondary Outcome: Number of Participants Who Experienced Mild Pain at Month 6 and 12: Tofacitinib Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 51
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 256 | 258 | 186 | 191
Participants | 44 | 40 | 28 | 25
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.55 to 1.46]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.47 to 1.51]

55. Secondary Outcome: Number of Participants Who Experienced Mild Pain at Month 6 and 12: Tofacitinib Combination Therapy Versus TNFi Combination Therapy
Description: as for outcome 51
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12 Month Follow-up)
Number analyzed (Participants) | 348 | 348 | 265 | 265
Participants | 62 | 56 | 39 | 36
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.60 to 1.38]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12 Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.56 to 1.50]

56. Secondary Outcome: Fatigue VAS at Month 6 and 12: Tofacitinib Overall Versus TNFi Overall
Description: Participants assessed their fatigue using a 0 to 100 mm VAS scale, where 0 mm = no fatigue and 100 mm = worst possible fatigue. Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 735 | 735 | 611 | 611
Millimeter | 46.23 (29.42) | 48.52 (30.19) | 46.75 (30.71) | 46.93 (29.83)
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 1.71, 95% CI 2-sided [-0.69 to 4.11]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-2.79 to 2.77]

57. Secondary Outcome: Fatigue VAS at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: as for outcome 56
Time Frame: Months 6 and 12 visit (for respective arms) post initiation of Tofacitinib during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 345 | 345 | 277 | 277
Millimeter | 48.31 (29.28) | 45.40 (29.33) | 48.51 (29.97) | 48.64 (31.20)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-5.02 to 1.60]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [-2.85 to 4.96]

58. Secondary Outcome: Fatigue VAS at Month 6 and 12: TNFi Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 56
Time Frame: Months 6 and 12 visit(for respective arms) post initiation of TNFis, during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 670 | 670 | 536 | 536
Millimeter | 46.25 (30.88) | 44.79 (29.48) | 46.20 (29.80) | 46.52 (30.31)
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-3.75 to 1.45]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Median Difference (Final Values) = -0.53, 95% CI 2-sided [-3.54 to 2.47]

59. Secondary Outcome: Fatigue VAS at Month 6 and 12: Tofacitinib Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 56
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 343 | 343 | 246 | 246
Millimeter | 47.11 (29.08) | 48.74 (28.89) | 48.90 (29.51) | 47.01 (30.62)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-2.36 to 4.73]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -3.15, 95% CI 2-sided [-7.36 to 1.07]

60. Secondary Outcome: Fatigue VAS at Month 6 and 12: Tofacitinib Combination Therapy Versus TNFi Combination Therapy
Description: as for outcome 56
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 443 | 443 | 344 | 344
Millimeter | 45.06 (29.00) | 48.02 (29.41) | 46.75 (31.10) | 47.62 (30.17)
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 2.37, 95% CI 2-sided [-0.66 to 5.41]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [-2.69 to 4.71]

61. Secondary Outcome: Morning Stiffness Duration at Month 6 and 12: Tofacitinib Overall Versus TNFi Overall
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in hours. Propensity score method was used for analysis of the outcome measure.
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tofacitinib Overall (6-Month Follow-up) | TNFis Overall (6-Month Follow-up) | Tofacitinib Overall (12-Month Follow-up) | TNFis Overall (12-Month Follow-up)
Number analyzed (Participants) | 735 | 735 | 611 | 611
Hours | 1.39 (2.73) | 1.56 (3.07) | 1.39 (2.96) | 1.51 (3.26)
Statistical Analysis 1: Comparison: Tofacitinib Overall (6-Month Follow-up) vs TNFis Overall (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.16 to 0.40]
Statistical Analysis 2: Comparison: Tofacitinib Overall (12-Month Follow-up) vs TNFis Overall (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.21 to 0.45]

62. Secondary Outcome: Morning Stiffness Duration at Month 6 and 12: Tofacitinib Monotherapy Versus Tofacitinib Combination Therapy
Description: as for outcome 61
Time Frame: as for outcome 57
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | Tofacitinib Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 345 | 345 | 277 | 277
Hours | 1.38 (2.60) | 1.48 (2.99) | 1.62 (3.24) | 1.41 (3.05)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs Tofacitinib Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.40 to 0.43]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs Tofacitinib Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.74 to 0.29]

63. Secondary Outcome: Morning Stiffness Duration at Month 6 and 12: TNFi Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 61
Time Frame: Months 6 and 12 visit (for respective arms) post initiation of TNFis during observation period from 06-November-2012 to 28-Feb-2021(approximately 8.3 years); data was collected and studied from 22-January-2021 to 29-November-2021 in this study
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | TNFis Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | TNFis Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 670 | 670 | 670 | 670
Hours | 1.51 (3.12) | 1.41 (2.74) | 1.49 (3.30) | 1.48 (2.95)
Statistical Analysis 1: Comparison: TNFis Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.51 to 0.10]
Statistical Analysis 2: Comparison: TNFis Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.42 to 0.31]

64. Secondary Outcome: Morning Stiffness Duration at Month 6 and 12: Tofacitinib Monotherapy Versus TNFi Combination Therapy
Description: as for outcome 61
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tofacitinib Monotherapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Monotherapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 343 | 343 | 246 | 246
Hours | 1.29 (2.30) | 1.28 (2.38) | 1.51 (3.08) | 1.53 (3.39)
Statistical Analysis 1: Comparison: Tofacitinib Monotherapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.34 to 0.32]
Statistical Analysis 2: Comparison: Tofacitinib Monotherapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.69 to 0.31]

65. Secondary Outcome: Morning Stiffness Duration at Month 6 and 12: Tofacitinib Combination Therapy Versus TNFi Combination Therapy
Description: as for outcome 61
Time Frame: as for outcome 11
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tofacitinib Combination Therapy (6-Month Follow-up) | TNFis Combination Therapy (6-Month Follow-up) | Tofacitinib Combination Therapy (12-Month Follow-up) | TNFis Combination Therapy (12-Month Follow-up)
Number analyzed (Participants) | 443 | 443 | 344 | 344
Hours | 1.41 (2.69) | 1.46 (2.95) | 1.39 (3.06) | 1.62 (3.46)
Statistical Analysis 1: Comparison: Tofacitinib Combination Therapy (6-Month Follow-up) vs TNFis Combination Therapy (6-Month Follow-up); Month 6 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.37 to 0.32]
Statistical Analysis 2: Comparison: Tofacitinib Combination Therapy (12-Month Follow-up) vs TNFis Combination Therapy (12-Month Follow-up); Month 12 follow-up visit analysis; Test type: Superiority; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.30 to 0.59]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not planned to be collected during the study
Description: Minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not collected and reported.
Groups:
- Tofacitinib (6 Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
- TNFis (6 Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) after 06-November-2012 and had at least 6-month follow-up post initiation, were included in this reporting arm.
- Tofacitinib (12 Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated tofacitinib after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
- TNFis (12 Month Follow-up): Participants diagnosed with RA, enrolled in Coronna RA registry who initiated TNFis (adalimumab, etanercept, infliximab, golimumab, or certolizumab pegol) after 06-November-2012 and had at least 12-month follow-up post initiation, were included in this reporting arm.
Arm/Group | Tofacitinib (6 Month Follow-up) | TNFis (6 Month Follow-up) | Tofacitinib (12 Month Follow-up) | TNFis (12 Month Follow-up)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04721821/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT04721821/SAP_001.pdf